CLINICAL TRIAL: NCT04838314
Title: Does Bilateral Continuous Peri Operative Erector Spinae Plane (ESP) Block Improve Analgesia and Reduce Opioid Consumption for Liver Transplantation in Recipient Paediatric Patient
Brief Title: Perioperative Analgesia by ESP Catheter on Paediatric Recipient for Liver Transplantation
Acronym: ESPLIVPAED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No More recruitment surgeon left the team
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VINMEC-LT-REC-PAED
Record Dates: First submitted 2021-04-01; First posted 2021-04-09 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Liver Transplant Disorder

STUDY DESIGN:
Intervention Model Description: randomized controlled prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of cares (No Intervention): Peri operative analgesia by opioids
- regional analgesia (Experimental): Peri operative analgesia by continuous bilateral ESP catheters
  Interventions: Procedure: regional analgesia

INTERVENTIONS:
Procedure: regional analgesia — Peri operative regional analgesia by bilateral ESP catheter for 72h
  Arms: regional analgesia

SUMMARY:
Pediatric Liver transplantation surgery is associated with moderate to severe postoperative pain that is related to large abdominal incision cutting muscles and fascia and the anterior abdominal wall and drains. Peri-operative pain management after this surgery is centered on intravenous opioids, which cannot provide complete pain relief and are responsible for side effects such as vomiting or respiratory depression. Fifty-two per cent of pediatric patients reported moderate to severe pain on the day of surgery and 33% on day 1. 42% of patients reported vomiting. Increasing interest has focused on opioid sparing analgesic strategies to avoid some of the detrimental side effects of opioids. Recently, the focus has been on postoperative regional analgesia after major pediatric in major thoracic or abdominal surgeries. Thoracic epidural anesthesia or paravertebral blocks are efficacious but raise some concerns related to their potential complications especially in Liver transplantation with the risk of coagulation disorders.

Erector spinae plane block (ESPB) is an interfascial plane block whereby Local anesthestic (LA) is injected beneath the iliocostalis, longissimus, and spinalis muscles to achieve multi metameric analgesia for pediatric thoracic, cardiac, or abdominal surgery.

I Investigators' hypothesis is with efficient peri operative regional analgesia will reduce the opioids consumption, allow a very early extubation after such long surgeries and improve the quality of recovery by reducing the side effects of opioids as sedation. nausea vomiting delay of first intake.

DETAILED DESCRIPTION:
1. Goals:

   Compare quality of analgesia and quality of recovery between bilateral ESP bilateral catheters versus Opioid analgesia in paediatric patients for liver transplantation reduce the peri operative opioid consumption
2. Methodology:

   * Selection criteria:

     * Age > 1 to 15 years old
     * Have a clinical indication for Liver transplantation ( list for surgeries listed in full proposal)
     * Agree to participate in the trial ( Parents or guardians)
   * Exclusion criteria:

     * Refusal participation.
     * Allergy to LA
     * Intubated ventilated pre-operation
     * Severe coagulation disorder
     * Coma
     * Prediction of large volume liver implanted
     * After surgery performed

       * Large volume implanted with a need of post operative controlled ventilation
       * Organ failure
     * Unstable patient
   * Study design: Prospective Randomized Controlled Trial.

   Patients who agree to join the study will be randomized into 2 groups:

   Group 1 (Control group): standard of care in Liver Transplantation for paediatric recipients: Intra-operative analgesia by Opioid sufentanil and post operative analgesia by patient controled analgesia assisted by nurse opioid morphine based on the protocol established by Prof Lee Vinmec transplantation surgical committee Group 2 (treatment group): Standard peri-operative analgesia for paediatric recipients in institution since we use regional anaesthesia as first line treatment for peri-operative analgesia Bilateral ESP catheters with continuous regional analgesia by infusion of local anesthestic (Ropivacaine) based on the guidelines by paediatric society of anesthesiologists and based on our recent article published in regional anaesthesia and pain medicine

   Sample size: We expected to reduce the peri operative opioid consumption by 85% for liver receipt The sample size of 10 patients per group is required to detect such changes assuming a confidence interval of 95% with a power of 90% and alpha = 0.05. Considering 20% of drop-out, the total sample size is 40 patients (20 patients each group)
3. Project outcomes:

The Primary outcome correlation between

* Pain quality evaluated by
* Opioids consumption The secondary outcomes
* Time to extubate
* Time to discharge from Intensive care Unit (ICU) we will create criteria to determinate when patient will discharge from ICU to go to high dependency In most of advanced hospital they don't keep a long time patient in ICU and send the patient to high dependency unit in surgery As in Institution we don't have we will keep the patient in ICU
* Time to discharge from hospital
* Time to first intake
* Any complication related to one type of analgesia

ELIGIBILITY:
Inclusion Criteria:

* Recipient liver transplantation who accepted to participate ( parents or guardians)

Exclusion Criteria:

* Refusal participation.
* Allergy to LA
* Intubated ventilated pre-operation
* Severe coagulation disorder
* Coma
* Prediction of large volume liver implanted
* After surgery performed Large volume implanted with a need of post operative controlled ventilation
* After surgery performed Organ failure
* After surgery performed Unstable patient

Ages: 12 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
peri operative Opioids consumption | up to day 7 after the end of surgery
  Dose of opioids used

SECONDARY OUTCOMES:
Time to extubate | up to 6 hours after the end of the surgery
  Time to reach the criteria to extubate after the end of the surgery
Duration of stay in Intensive care Unit (ICU) | up to 72 hours after the end of the surgery
  Time to reach the criteria of ICU discharge after liver transplantation
Length of stay in hospital | up to 30 day after the end of the surgery
  Time to reach the criteria of hospital discharge after liver transplantation
first intake | up to 72hours after the end of the surgery
  Time to have first intake after the end of the surgery
first mobilisation | up to 72hours after the end of the surgery
  Time to have first stand up after the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: philippe Macaire, MD, Principal Investigator — VinMEC
Locations (1):
- VinMec International hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No